CLINICAL TRIAL: NCT00414856
Title: A Multi-Center, Randomized, Double-Blind, Placebo- and Positive-Control, Double-Dummy, 3 Parallel Cohort, Two-Way Crossover Single Oral Dose Study in GERD (Gastro Esophageal Reflux Disease) Patients to Evaluate the Effects of AFQ056 and Baclofen (Positive Control) on the Incidence of Meal-Induced Gastro Esophageal Reflux Events
Brief Title: Effects of AFQ056 and Baclofen on Meal-Induced Gastroesophageal Reflux
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CAFQ056A2108
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; gastroesophageal reflux disease; meal-induced gastroesophageal reflux events
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — mavoglurant

INTERVENTIONS:
Drug: AFQ056

SUMMARY:
This study will assess the safety and tolerability of oral single dose applications of AFQ056 in GERD patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with GERD (18-60 years) with a history of moderate to severe reflux symptoms (heartburn or acid regurgitation more than 2 days/week, and/or night-time reflux, and/or after meal reflux) for ≥ 3 months with:

  * uncomplicated reflux-esophagitis of any degree as evidenced by esophagogastroduodenoscopy (EGD) within the last 12 months, OR (and) a pathological ambulatory 24-hours pH measurement within the last 12 months with pH < 4 for ≥ 9% of the time.
* Females must be of no child bearing potential (postmenopausal women with no regular menstrual bleeding for at least 1 year or women who have been surgically sterilized at least 6 months prior). Menopause will be confirmed by a plasma FSH level of 37.0 - 185.0 mIU/mL. Surgical sterilization procedures must be supported with clinical documentation.
* Patients must be able to completely finish the high-fat breakfast within 15 minutes.
* Body mass index must be below 30. Patients must weigh at least 60 kg to participate in this study.
* Patients must be able to communicate well with the investigator, to understand and comply with the requirements of the study and to understand and sign the written informed consent.

Exclusion Criteria:

History of:

* Upper gastrointestinal (GI) surgery or radiation
* GI disorders other than GERD that may significantly affect the incidence and/or assessment of reflux episodes (GI motility disorders, connective tissue disease like scleroderma, Barrett's esophagus, hiatal hernia > 3-4 cm, previous esophageal bleeding, esophageal varices, active gastric or duodenal ulcer disease, active esophagitis
* Delayed gastric emptying, or endoscopic indications for a delay in gastric emptying or gastric outlet obstruction.
* Neurologic/psychiatric disorders including a family history of epilepsy clinically significant cardiac disease
* Diabetes mellitus or other metabolic disorders including hyperlipidemia requiring treatment
* Any significant acute or chronic conditions except for following treated by the quoted drugs with a stable therapy for at least 4 weeks:

  * Hypertension well-controlled with the following:

    1. ACE inhibitors: benazepril, captopril, cilazapril, enalapril, fosinopril, imidapril, lisinopril, moexipril, perindopril tert-butylamine, quinapril, ramipril, spirapril, trandolapril, zofenopril, and/or
    2. angiotensin II receptor antagonists: candesartan cilexetil, eprosartan, irbesartan, losartan, olmesartan, telmisartan, valsartan, and/or
    3. diuretics: amiloride, bendroflumethiazide, bumetanide, canrenoate de potassium, chlortalidone, cicletanine, clopamide, cyclothiazide, furosemide, hydrochlorothiazide, indapamide, methyclothiazide, piretanide, spironolactone, torasemide, triamterene, xipamide, and/or
    4. calcium antagonists: bepridil, felodipine, isradipine, lercanidipine, manidipine, nimodipine, nitrendipine, amlodipine, nicardipine BUT NOT diltiazem, nifedipine, verapamil
  * Well-compensated asthma with topical use of corticosteroids and/or β2-mimetics
  * Patients on thyroid hormone therapy with a normal TSH value.
* Nonsteroidal anti-inflammatory drugs including aspirin use in the week prior to treatment/impedance monitoring.
* Patients with body mass index ≥ 30.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2006-08

PRIMARY OUTCOMES:
Gastroesophageal reflux episodes as assessed by impedance measurements in the 4-hour period following a standardized high-fat meal in patients with GERD.

SECONDARY OUTCOMES:
Safety and tolerability of oral AFQ056 in GERD patients.
Pharmacokinetics (PK) of two AFQ056 single oral doses in patients with GERD.
Relationships between AFQ056 blood levels and/or how the body interacts with the medication and overall reflux incidence
Validation of the reflux model used in this study using baclofen as positive control.
Effects of AFQ056 on other impedance/pH parameters, including but not limited to the rate of reflux episodes at various time intervals

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (4):
- Novartis Investigative site, Brussels, Belgium
- Novartis Investigative site, Paris, France
- Novartis Investigative Site, Nuremberg, Germany
- Novartis Investigative site, Bern, Switzerland